CLINICAL TRIAL: NCT05669924
Title: The Neural Correlates of and Effects of Methylphenidate on Acute Pain Dynamics
Brief Title: Neural Correlates of Acute Pain Dynamics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Andrew Vigotsky, PhD Candidate, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU00213557
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: Mesolimbic system; Dopamine circuits; Psychophysics
MeSH Terms: conditions — Pain | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — 0.35 mg/kg methylphenidate will be administered after baseline testing and 45 min-1 hr before post-intervention testing.
  Arms: Methylphenidate
Drug: Placebo — Placebo for methylphenidate
  Arms: Placebo

SUMMARY:
This work aims to study the neural correlates and determinants of pain dynamics related to changes in a noxious stimulus.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Pregnant
* History of chronic pain
* History of neurological diagnosis
* History of psychiatric diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Effect of methylphenidate on acute pain dynamics | 6 months
  We will compare acute pain dynamics-i.e., the time series of pain visual analog scale ratings (0-100, where 0 = no pain and 100 = worst pain imaginable) obtained while delivering a changing noxious stimulus-during the methylphenidate condition to that of the placebo condition.
Nucleus accumbens activation with acute pain dynamics | 6 months
  We will regress the time course of nucleus accumbens BOLD activity onto the latent time series obtained from our valence competition model. This will be supported by regressing the nucleus accumbens time course onto the pain VAS time course, allowing our findings to be compared to standard analyses in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Vigotsky, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized and shared on OpenPain.org upon publication.
Supporting Information: Analytic Code
Time Frame: 1 year